CLINICAL TRIAL: NCT06899230
Title: A Phase 1, Randomized, Double-blind, Placebo-controlled, Single and Multiple Ascending Dose Study to Assess the Safety, Tolerability and Pharmacokinetics of Oral iQ-007 in Healthy Male and Female Adult Participants
Brief Title: Safety, Tolerability, and Pharmacokinetics (PK) of Single and Multiple Ascending Oral Doses of iQ-007
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: iQure Australia Pty Ltd (Industry)
Collaborators: Avance Clinical Pty Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: iQ-007-CL-001
Record Dates: First submitted 2025-03-13; First posted 2025-03-27 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Drug Resistant Epilepsy; Focal Seizure
MeSH Terms: conditions — Drug Resistant Epilepsy; Seizures

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- iQ-007 (Experimental): Part A (SAD): a total of 48 healthy volunteers are planned to be enrolled across 6 SAD cohorts and will involve the administration of a single oral dose of iQ-007 (in the range of 200 mg up to 2800 mg) or placebo capsules on Day 1.
  Part B (MAD): a total of 24 healthy volunteers are planned to be enrolled across 3 MAD cohorts and will involve the administration of multiple twice daily oral doses of iQ-007 (in the range of 600 mg up to 2400mg total per day) or placebo capsules on Days 1 to 14.
  Interventions: Drug: iQ-007
- Placebo (Placebo Comparator): Part A (SAD): a total of 48 healthy volunteers are planned to be enrolled across 6 SAD cohorts and will involve the administration of a single oral dose of iQ-007 (in the range of 200 mg up to 2800 mg) or placebo capsules on Day 1.
  Part B (MAD): a total of 24 healthy volunteers are planned to be enrolled across 3 MAD cohorts and will involve the administration of multiple twice daily oral doses of iQ-007 (in the range of 600 mg up to 2400mg total per day) or placebo capsules on Days 1 to 14.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: iQ-007 — Highly selective, orally bioavailable, positive allosteric modulator (PAM) of the excitatory amino acid transporter-2 (EAAT2) and its rodent homologue (glutamate transporter-1[GLT-1).
  Arms: iQ-007
Drug: Placebo — Oral capsules identical in appearance to drug and containing vehicle only (Gelucire/Capmul-M).
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled study conducted in healthy adult volunteers to assess the safety, tolerability and pharmacokinetics of iQ-007. iQ-007 may be indicated for use in patients with Focal Seizures and Drug-resistant Epilepsy (DRE).

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled study conducted in healthy adult volunteers. The study will be conducted in 2 parts: a single ascending dose (SAD) component and a multiple ascending dose (MAD) component.

Part A (SAD) will involve the administration of a single oral dose of iQ-007 or placebo capsules on Day 1 in Cohorts Al, A2, A3, A5 and A6. Participants in Cohort A4, will be required to fast overnight (minimum of 8 hours) prior to eating a high fat breakfast 30 minutes prior to a single oral administration of iQ-007 or placebo capsules on Day 1.

Part B (MAD) will involve the administration of multiple twice daily oral doses of iQ-007 or placebo capsules on Days 1 to 14 (total of 27 doses) in cohorts B1, B2, B3.

ELIGIBILITY:
Inclusion Criteria:

1. Must have given written informed consent before any study-related activities are performed and must be able to understand the full nature and purpose of the study, including possible risks and adverse effects.
2. Adult males or females, 18 to 55 years of age (inclusive) at screening.
3. Body mass index (BMI) greater than or equal to 18.0 and less than or equal to 32.0 kg/m2.
4. Medically healthy (in the opinion of the PI), as determined by pre-study medical history, and without clinically significant (CS) abnormalities including the following:

   1. Physical examination without any clinically relevant findings.
   2. Systolic blood pressure in the range of 90 to 160 mmHg and diastolic blood pressure in the range of 50 to 95 mmHg after resting for 5 minutes in a supine or semi-supine position.
   3. Pulse rate in the range of 45 to 100 bpm after 5 minutes resting in a supine or semi-supine position.
   4. Body temperature (tympanic), between 35.5°C and 37.7°C. If temperature above 36.6°C, any infective etiology must be ruled out by the PI.
   5. Electrocardiogram without CS abnormalities including QT interval corrected for Fredericia (QTcF) <450msec
   6. No CS findings in serum chemistry, hematology, coagulation, and urinalysis tests.
5. Female volunteers:

   1. Must be of non-childbearing potential, i.e., surgically sterilized (hysterectomy, bilateral salpingectomy, bilateral oophorectomy) at least 6 weeks before the screening visit or postmenopausal (where postmenopausal is defined as no menses for 12 months without an alternative medical cause and a follicle-stimulating hormone [FSH] level consistent with postmenopausal status, per local laboratory guidelines), or
   2. If of childbearing potential, must:

   i. Have a negative pregnancy test at the screening visit and on admission to the study site on Day-1.

   ii. Agree not to attempt to become pregnant or donate ova from signing the consent form until at least 90 days after the last dose of the study drug.

   iii. Agree to use adequate contraception (defined as use of a condom by the male partner combined with use of a highly effective method of contraception) established at screening until at least 30 days after the last dose of the study drug, if not exclusively in a same-sex relationship, or in relationship without a risk of pregnancy (sterile partner), or abstinent as a committed lifestyle.
6. Male volunteers, must:

   1. Agree not to donate sperm from signing the consent form until at least 90 days after the last dose of the study drug.
   2. If engaging in sexual intercourse with a female partner who could become pregnant, agree to use adequate contraception (defined as use of a condom combined with their female partner's use of a highly effective method of contraception) from signing the consent form until at least 90 days after the last dose of the study drug.
   3. If engaging in sexual intercourse with a partner who is not at risk of pregnancy (sterile partner), agree to use a condom from signing the consent form until at least 90 days after the last dose of the study drug.
7. For SAD Cohort A4 only: Willing and able to adhere to standard high fat, high calorie meal.
8. Have suitable venous access for blood sampling.
9. Willing and able to comply with all study assessments and adhere to the protocol schedule and restrictions.

Exclusion Criteria:

1. Known hypersensitivity to any of the study drug ingredients.
2. History of anaphylaxis or other significant allergy which, in the opinion of the PI, would interfere with the volunteer's ability to participate in the study.
3. History or presence of CS cardiovascular, pulmonary, hepatic, renal, hematological, gastrointestinal/bariatric modification, endocrine, immunologic, dermatologic, psychiatric, or neurological disease/disorder, including any acute illness, within the past 3 months determined by the PI to be clinically relevant.

   Note: Participants with history of resolved childhood asthma, psoriasis, atopic dermatitis, non-hospitalized depression, anxiety and/or migraine are permitted to be included in the study.
4. History of surgery or hospitalization within 3 months prior to screening, or elective surgery planned during the study.
5. Any history of malignant disease in the last 10 years (excludes surgically resected skin squamous cell or basal cell carcinoma).
6. Presence of clinically relevant immunosuppression from, but not limited to, immunodeficiency conditions such as common variable hypogammaglobulinemia.
7. History of risk factors for torsade de pointes (including a family history of long QT syndrome or sudden cardiac death) or a known arrythmia.
8. Presence or having sequelae of gastrointestinal, liver (including Gilbert's syndrome), kidney, or other conditions known to interfere with the absorption, distribution, metabolism, or excretion of drugs.
9. Liver function test results elevated >1.5-fold above the ULN for gamma glutamyl transferase, bilirubin(total), ALP, AST or ALT. Volunteers with ALP and/or ALT/AST above the limits specified may be included, at the discretion of the PI (or delegate), if the levels are unaccompanied by clinical signs and are determined to be normal variants.
10. Estimated creatinine clearance <60 mL/min using the Cockcroft-Gault formula or serum creatinine>1.2-fold above the ULN.
11. A history of or positive test results for human immunodeficiency virus (HIV), hepatitis B surface antigen(HBsAg) or hepatitis C (HCV) at the screening visit. Note that a history of hepatitis C virus (HCV) is not exclusionary and if deemed cured by the PI, may be included on a case-by-case basis at the MM and Sponsor's discretion.
12. Positive drugs of abuse test, cotinine test or alcohol breath test results at the screening visit and/or on admission to the study site on Day -1.
13. Regular consumption of more than 10 standard alcoholic drinks/week and/or more than 4 standard alcoholic drinks on any one day, where 1 standard drink is 10 g of pure alcohol and is equivalent to 285 mL beer [4.9% Alc/Vol], 100 mL wine [12% Alc/Vol], or 30 mL spirit [40% Alc/Vol]).
14. Volunteer smokes more than 5 cigarettes or equivalent nicotine-containing products per week, and/or the volunteer is unwilling to abstain from smoking or the use of nicotine-containing products for 72 hours prior to check-in on Day -1 and throughout the confinement period at the study site.
15. Females who are breastfeeding or planning to breastfeed.
16. Unable to swallow oral medication.
17. Use of any prescription or over-the-counter medication (including herbal products, diet aids, vitamins, and hormone supplements) within 10 days or 5 half-lives of the medication (whichever is longer) prior to the first dose of study drug, except use of contraceptives, the use of paracetamol (up to 2 g per day) for over 3 consecutive days and the use of ibuprofen (up to 1.2 g per day) for over 3 consecutive days.
18. Current infection that requires systemically absorbed antibiotic, antifungal, antiparasitic or antiviral medication within 10 days prior to first dose of study drug.
19. Use of any vaccinations within 30 days prior to screening.
20. Donation of blood or plasma within 30 days prior to first dose of study drug, or loss of whole blood of more than 500 mL within 30 days prior to first dose of study drug, or receipt of a blood transfusion within 1year of the first dose of study drug.
21. Participation in any clinical study of an investigational drug or investigational device within 30 days or 5 half-lives of the investigational drug (whichever is longer) prior to screening.
22. Any other condition or prior therapy that in the opinion of the PI (or delegate) would make the volunteer unsuitable for this study, including inability to cooperate fully with the requirements of the study protocol or likelihood of noncompliance with any study requirements.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Estimated)
Dates: Start 2025-04-08 (Actual); Primary Completion 2026-01-29 (Estimated); Study Completion 2026-01-29 (Estimated)

PRIMARY OUTCOMES:
Incidence, severity and relationship of treatment-emergent adverse events (TEAEs), serious adverse events (SAEs), and TEAEs. | From baseline to the end of observation on Day 8 for Single ascending dose. From baseline to the end of observation on Day 21 for Multiple ascending dose.
  Adverse event (AE) - graded using the categories Mild, Moderate or Severe and will be classified as normal, abnormal not clinically significant (NCS), or abnormal CS.
Changes from baseline in Blood pressure measurements | From baseline to the end of observation on Day 8 for Single ascending dose. From baseline to the end of observation on Day 21 for Multiple ascending dose.
  Vital signs assessed as normal, abnormal not clinically significant (NCS), or abnormal clinically significant (CS) with Blood pressure assessed using digital sphygmomanometer
Changes from baseline in electrocardiogram (ECG) parameters | From baseline to the end of observation on Day 8 for Single ascending dose. From baseline to the end of observation on Day 21 for Multiple ascending dose.
  Twelve-lead Electrocardiogram's (ECG's) including the measurement of ventricular heart rate [HR] will be conducted in triplicate.
Changes from baseline in clinical laboratory results | From baseline to the end of observation on Day 8 for Single ascending dose. From baseline to the end of observation on Day 21 for Multiple ascending dose.
  Clinical laboratory results assessed using blood and urine samples and will be classified as normal, abnormal not clinically significant (NCS), or abnormal CS.
Changes from baseline in heart rate measurements | From baseline to the end of observation on Day 8 for Single ascending dose. From baseline to the end of observation on Day 21 for Multiple ascending dose.
  Vital signs assessed as normal, abnormal not clinically significant (NCS), or abnormal CS with heart rate and respiratory rate assessed using pulse oximeter
Changes from baseline in temperature measurements | From baseline to the end of observation on Day 8 for Single ascending dose. From baseline to the end of observation on Day 21 for Multiple ascending dose.
  Vital signs assessed as normal, abnormal not clinically significant (NCS), or abnormal CS with temperature assessed using digital thermometer.
Changes from baseline in ECG PR interval | From baseline to the end of observation on Day 8 for Single ascending dose. From baseline to the end of observation on Day 21 for Multiple ascending dose.
  Twelve-lead Electrocardiogram's (ECG's) including the measurement of PR interval will be conducted in triplicate.
Changes from baseline in ECG QRS duration | From baseline to the end of observation on Day 8 for Single ascending dose. From baseline to the end of observation on Day 21 for Multiple ascending dose.
  Twelve-lead Electrocardiogram's (ECG's) including the measurement of QRS duration will be conducted in triplicate.
Changes from baseline in ECG QT interval | From baseline to the end of observation on Day 8 for Single ascending dose. From baseline to the end of observation on Day 21 for Multiple ascending dose.
  Twelve-lead Electrocardiogram's (ECG's) including the measurement of QT interval will be conducted in triplicate.
Changes from baseline in ECG QTcF | From baseline to the end of observation on Day 8 for Single ascending dose. From baseline to the end of observation on Day 21 for Multiple ascending dose.
  Twelve-lead Electrocardiogram's (ECG's) including the measurement of QTcF will be conducted in triplicate.

SECONDARY OUTCOMES:
Single Ascending Dose: Plasma PK parameter - Maximum observed concentration (Cmax) | Pre-dose Day 1, then 0.5, 1, 2, 3, 4, 6, 8, 12 and 16 hours post-dose, Day 2, 24 hours post-dose, Day 3, 48 hours post-dose, Day 4, 72 hours post-dose and Day 5, 96 hours post-dose.
  Blood plasma samples will be assessed
Multiple Ascending Dose: Plasma PK parameters - Maximum observed concentration (Cmax) | pre-dose Day 1 then 0.5, 1, 2, 3, 4, 6, 8, & 12 hrs post-dose, pre-dose on Days 2 - 13, pre-dose Day 14 then 0.5, 1, 2, 3, 4, 6, 8, 12 & 16 hrs post-dose, Day 15 24 hrs post-dose, Day 16 48 hrs post-dose, Day 17 72 hrs post-dose & Day 18 96 hrs post-dose
  Blood plasma samples will be assessed
Multiple ascending dose: Urine PK endpoints include • Cumulative amount of un-changed drug excreted inurine (Ae) | Pre-dose Day 1 - up to 12 hours post AM (first) dose, Day 14 and Day 15, up to 12 hours post AM (final) dose, 12 to 24 hours post AM (final) dose, Day 16, 24 to 48 hours post-dose, Day 17, 48 to 72 hours post-dose and Day 18, 72 to 96 hours post-dose.
  Urine samples will be assessed
Single Ascending Dose: Plasma PK parameter - Time to maximum observed concentration (Tmax) | Pre-dose Day 1, then 0.5, 1, 2, 3, 4, 6, 8, 12 and 16 hours post-dose, Day 2, 24 hours post-dose, Day 3, 48 hours post-dose, Day 4, 72 hours post-dose and Day 5, 96 hours post-dose.
  Blood plasma samples will be assessed
Single Ascending Dose: Plasma PK parameter - Area under the concentration-time curve from 0 to time of last quantifiable concentration (AUClast) | Pre-dose Day 1, then 0.5, 1, 2, 3, 4, 6, 8, 12 and 16 hours post-dose, Day 2, 24 hours post-dose, Day 3, 48 hours post-dose, Day 4, 72 hours post-dose and Day 5, 96 hours post-dose.
  Blood plasma samples will be assessed
Single Ascending Dose: Plasma PK parameter - Area under the concentration-time curve from time 0 extrapolated to infinity (AUCinf) | Pre-dose Day 1, then 0.5, 1, 2, 3, 4, 6, 8, 12 and 16 hours post-dose, Day 2, 24 hours post-dose, Day 3, 48 hours post-dose, Day 4, 72 hours post-dose and Day 5, 96 hours post-dose.
  Blood plasma samples will be assessed
Single Ascending Dose: Plasma PK parameter - Apparent terminal elimination half-life (T1/2) | Pre-dose Day 1, then 0.5, 1, 2, 3, 4, 6, 8, 12 and 16 hours post-dose, Day 2, 24 hours post-dose, Day 3, 48 hours post-dose, Day 4, 72 hours post-dose and Day 5, 96 hours post-dose.
  Blood plasma samples will be assessed
Single Ascending Dose: Plasma PK parameter - Volume of distribution (Vz/F) | Pre-dose Day 1, then 0.5, 1, 2, 3, 4, 6, 8, 12 and 16 hours post-dose, Day 2, 24 hours post-dose, Day 3, 48 hours post-dose, Day 4, 72 hours post-dose and Day 5, 96 hours post-dose.
  Blood plasma samples will be assessed
Single Ascending Dose: Plasma PK parameter - Clearance (CL/F) | Pre-dose Day 1, then 0.5, 1, 2, 3, 4, 6, 8, 12 and 16 hours post-dose, Day 2, 24 hours post-dose, Day 3, 48 hours post-dose, Day 4, 72 hours post-dose and Day 5, 96 hours post-dose.
  Blood plasma samples will be assessed
Multiple Ascending Dose: Plasma PK parameters - Time to maximum observed concentration (Tmax) | Pre-dose Day 1 0.5, 1, 2, 3, 4, 6, 8, & 12 hours post-dose, pre-dose Days 2 - 13, pre-dose Day 14 0.5, 1, 2, 3, 4, 6, 8, 12 & 16 hours post-dose, Day 15 24 hours post-dose, Day 16 48 hours post-dose, Day 17 72 hours post-dose, Day 18 96 hours post-dose
  Blood plasma samples will be assessed
Multiple Ascending Dose: Plasma PK parameter - Area under the concentration-time curve from 0 to time of last quantifiable concentration (AUClast) | Pre-dose Day 1 0.5, 1, 2, 3, 4, 6, 8, & 12 hours post-dose, pre-dose Days 2 - 13, pre-dose Day 14 0.5, 1, 2, 3, 4, 6, 8, 12 & 16 hours post-dose, Day 15 24 hours post-dose, Day 16 48 hours post-dose, Day 17 72 hours post-dose, Day 18 96 hours post-dose
  Blood plasma samples will be assessed
Multiple Ascending Dose: Plasma PK parameter - Area under the concentration versus time curve for the dosing interval (AUCtau) | Pre-dose Day 1 0.5, 1, 2, 3, 4, 6, 8, & 12 hours post-dose, pre-dose Days 2 - 13, pre-dose Day 14 0.5, 1, 2, 3, 4, 6, 8, 12 & 16 hours post-dose, Day 15 24 hours post-dose, Day 16 48 hours post-dose, Day 17 72 hours post-dose, Day 18 96 hours post-dose
  Blood plasma samples will be assessed
Multiple Ascending Dose: Plasma PK parameter - Area under the concentration-time curve from time 0 extrapolated to infinity (AUCinf) | Pre-dose Day 1 0.5, 1, 2, 3, 4, 6, 8, & 12 hours post-dose, pre-dose Days 2 - 13, pre-dose Day 14 0.5, 1, 2, 3, 4, 6, 8, 12 & 16 hours post-dose, Day 15 24 hours post-dose, Day 16 48 hours post-dose, Day 17 72 hours post-dose, Day 18 96 hours post-dose
  Blood plasma samples will be assessed
Multiple Ascending Dose: Plasma PK parameter - Apparent terminal elimination half-life (T1/2) | Pre-dose Day 1 0.5, 1, 2, 3, 4, 6, 8, & 12 hours post-dose, pre-dose Days 2 - 13, pre-dose Day 14 0.5, 1, 2, 3, 4, 6, 8, 12 & 16 hours post-dose, Day 15 24 hours post-dose, Day 16 48 hours post-dose, Day 17 72 hours post-dose, Day 18 96 hours post-dose
  Blood plasma samples will be assessed
Multiple Ascending Dose: Plasma PK parameter - Volume of distribution (Vz/F) | Pre-dose Day 1 0.5, 1, 2, 3, 4, 6, 8, & 12 hours post-dose, pre-dose Days 2 - 13, pre-dose Day 14 0.5, 1, 2, 3, 4, 6, 8, 12 & 16 hours post-dose, Day 15 24 hours post-dose, Day 16 48 hours post-dose, Day 17 72 hours post-dose, Day 18 96 hours post-dose
  Blood plasma samples will be assessed
Multiple Ascending Dose: Plasma PK parameter - Clearance (CL/F) | Pre-dose Day 1 0.5, 1, 2, 3, 4, 6, 8, & 12 hours post-dose, pre-dose Days 2 - 13, pre-dose Day 14 0.5, 1, 2, 3, 4, 6, 8, 12 & 16 hours post-dose, Day 15 24 hours post-dose, Day 16 48 hours post-dose, Day 17 72 hours post-dose, Day 18 96 hours post-dose
  Blood plasma samples will be assessed
Multiple Ascending Dose: Plasma PK parameter - Accumulation ratio for Maximum observed concentration (Cmax) and Area under the concentration versus time curve for the dosing interval (AUCtau) using the first and last dose | Pre-dose Day 1 0.5, 1, 2, 3, 4, 6, 8, & 12 hours post-dose, pre-dose Days 2 - 13, pre-dose Day 14 0.5, 1, 2, 3, 4, 6, 8, 12 & 16 hours post-dose, Day 15 24 hours post-dose, Day 16 48 hours post-dose, Day 17 72 hours post-dose, Day 18 96 hours post-dose
  Blood plasma samples will be assessed
Multiple ascending dose: Urine PK endpoints include • Fraction of the dose excreted in urine (Fe) | Pre-dose Day 1 - up to 12 hours post AM (first) dose, Day 14 and Day 15, up to 12 hours post AM (final) dose, 12 to 24 hours post AM (final) dose, Day 16, 24 to 48 hours post-dose, Day 17, 48 to 72 hours post-dose and Day 18, 72 to 96 hours post-dose.
  Urine samples will be assessed
Multiple ascending dose: Urine PK endpoints include • Renal clearance (CLr). | Pre-dose Day 1 - up to 12 hours post AM (first) dose, Day 14 and Day 15, up to 12 hours post AM (final) dose, 12 to 24 hours post AM (final) dose, Day 16, 24 to 48 hours post-dose, Day 17, 48 to 72 hours post-dose and Day 18, 72 to 96 hours post-dose.
  Urine samples will be assessed

CONTACTS AND LOCATIONS:
Overall Officials: Henk de Wilde, Study Director — iQure Australia Pty Ltd
Locations (1):
- CMAX Clinical Research Pty Ltd, Adelaide, South Australia, Australia

IPD SHARING:
Plan to Share IPD: No